CLINICAL TRIAL: NCT06145074
Title: Examining the Impact of Propranolol on Preoperative Anxiety and on Tumorigenic Changes in Patients With Pancreatic Ductal Adenocarcinomas: a Randomized, Triple-blinded, Placebo-controlled Pilot Trial
Brief Title: Examining Safety, Efficacy and Feasibility of Preoperative Propranolol in Patients With PDAC.
Acronym: IMPULS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EU CT 2023-506553-37-00
Record Dates: First submitted 2023-11-08; First posted 2023-11-22 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Cancer; Surgery
Keywords: Propranolol; Beta-Blockers; PDAC; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol (Experimental): Propranolol will be administered 40 mg twice daily (morning and evening) in 10 days prior to surgery for pancreatic cancer
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Placebo will be administered twice daily (morning and evening) in 10 days prior to surgery for pancreatic cancer.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Oral administration.
  Other Names: Inderal; Propal
  Arms: Propranolol
Drug: Placebo — Oral administration.
  Other Names: Inactive drug
  Arms: Placebo

SUMMARY:
The IMPULS trial is a randomized, triple-blinded, placebo controlled, single center, pilot trial examining the efficacy and safety of preoperative propranolol in patients scheduled for pancreatic cancer surgery. The study is conducted as a type 1 hybrid efficacy-implementation trial of 30 patients.

This study is designed to provide pilot data for a future larger perioperative study of propranolol with the aim of improving outcomes for pancreatic cancer surgery.

In total, 30 participants will be allocated in a 1:1 ratio with 15 participants enrolled in each trial arm (propranolol vs. placebo). Participants will be allocated to either 40 mg propranolol twice daily or placebo twice daily in 10 days prior to planned surgery.

Primary outcomes: Evaluating the efficacy of preoperative propranolol on anxiety and in pro-tumorigenic changes (e.g., in the tumor tissue and in blood samples) in patients undergoing surgery for pancreatic cancer. Furthermore, to obtain follow up data (e.g., 90-day mortality, postoperative complications etc. on the patients receiving propranolol versus placebo). Heart rate variability among the participants will also be examined.

Secondary: Examining the safety and tolerability of 40 mg preoperative propranolol twice daily in patients undergoing surgery for pancreatic cancer.

Tertiary: Evaluating the feasibility and implementation of the trial (using the APEASE framework). This will help identify barriers and enablers to a future larger study.

Short-time propranolol treatment is considered safe with a mild and manageable safety-profile. Risk-management, mitigations and guidelines to ensure patient safety is included in the protocol. Since this clinical trial is exploratory in nature, no sample-size calculation is performed.

DETAILED DESCRIPTION:
The study will be conducted as a pilot study to test efficacy, safety and feasibility of propranolol on preoperative anxiety in patients undergoing abdominal surgery for suspected pancreatic ductal adenocarcinoma (PDAC). Furthermore, the implementation of the trial including compliance of the participants in a hybrid type 1 setup will be examined.

A total of 30 participants will be included and randomized to receive either propranolol or placebo twice daily with 15 patients in each arm. Following this study, a power calculation will be done to reveal the actual number of needed participants in each arm for a potential follow-up randomized clinical trial on primary outcomes of interest. Thus, the results from this study can be used for future power calculations for clinical trials related to this topic.

Primary objectives: Efficacy

Evaluating the efficacy of preoperative propranolol on patient-experienced anxiety and on tumorigenic gene expression compared to placebo is the primary objective of this trial.

Primary objectives are further divided in to primary clinical objectives, primary translational objectives and exploratory endpoints.

Primary clinical objectives:

The primary clinical objectives are to evaluate preoperative patient-experienced anxiety in patients receiving the nonselective beta-2-adrenergic receptor inhibitor, propranolol, compared to placebo.

Further, heart rate variability (HRV) will be measured in order to evaluate changes in the autonomous nervous system in relation to surgery. HRV is calculated from the interval variation between consecutive R waves in an ECG time series and results suggest that it is associated with the intra- and postoperative complications. As HRV reflects sinoatrial node regulation, it is expected to be affected by the beta-adrenergic blockade caused by preoperative propranolol. Analyzing this relation will provide essential knowledge in understanding how HRV behaves perioperatively.

Lastly, follow up on the participants receiving propranolol compared to placebo will be done.

Primary clinical effect parameters:

The following primary effect parameters will be used to investigate the primary clinical objectives:

* Anxiety levels will primarily be measured by The Hamilton Anxiety Rating Scale (HAM-A) and secondarily by The Hospital Anxiety and Depression Scale (HADS). The European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QoL) for pancreatic cancer will be used to assess quality of life.
* HRV is calculated from continuous ECG gathered by a Holter monitor. The monitor is a small wearable apparatus with one lead, placed on the patient's sternum. It is applied on preoperative day 9 and will run continually until approximately postoperative day 7. The actual calculations are achieved post hoc using software specialized for HRV analysis.
* Follow up at 30- and 90-days after surgery including parameters such as survival and postoperative complications.
* Long-term follow up at as 1-year, 3- year and 5-year following surgery including survival and recurrence data.

Primary translational objectives:

The primary translational objectives are to examine the systemic (biochemical) and local changes (TME of resections) to propranolol treatment compared to placebo. Alterations in pro-metastatic and proinflammatory genes will specifically be analyzed.

Primary translational effect parameters:

* Blood sampling for the analysis of pro-metastatic and proinflammatory biomarkers.
* Expression of pro-metastatic and proinflammatory genes in formalin-fixed paraffin-embedded (FFPE) cancer tissue obtained after surgical resection.

Exploratory endpoints:

The potential influence of inter-participant genetic variations (pharmacogenetics) on measured levels of serum propranolol and response to surgical stress will be investigated as exploratory endpoints. The differences in drug metabolism (pharmacokinetics) among participants will also be of interest.

Secondary objectives: Safety

Secondarily, tolerance and safety of the intervention in this pilot study (e.g., adverse effects, number of patients that need dose reduction etc.) will be evaluated. Changes in heart rate (HR) and blood pressure (BP) during the intervention period will be examined to test safety and tolerability of preoperative propranolol.

Secondary effect parameters:

* Measuring the changes in resting HR and BP during the intervention period with handed out blood pressure monitors.
* Safety endpoints: light-headedness, lethargy, hypotension, bradycardia and other symptoms and side-effects that may be related to propranolol treatment.

Tertiary objectives: Feasibility

Additionally, the feasibility of this intervention using the APEASE framework, which assesses factors like affordability, practicability, effectiveness, acceptability, side-effects, and equity, thereby determining the willingness to adopt this strategy will be examined. This will help identify barriers and enablers to a future larger study. The details regarding the APEASE framework are described under assessments.

This trial will be conducted in accordance with the principles of Good Clinical Practice and reported according to the CONSORT and the complimentary StaRI standards for implementation studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected surgically resectable pancreatic cancer
* Indication for surgical treatment with curative intend.
* Provide written informed consent.
* Patients minimum 18 years old.

Women of childbearing potential (WOCBP) are defined as women ranging from the period of menarche till the post-menopausal period, unless permanently sterile (e.g., hysterectomy, bilateral salpingectomy and bilateral oophorectomy). Post-menopause is defined as no menses for 12 months without an alternative medical cause.

WOCBP should use a secure and highly effective birth control (as stated in the "Recommendations related to contraception and pregnancy testing in clinical trials", version 1.1., section 4.1, from the Clinical Trials Facilitation and Coordination Group) during the entire period of the trial. In cases of uncertainty regarding pregnancy, additional pregnancy testing either as highly sensitive serum or urine pregnancy test can be used.

Exclusion Criteria:

* Patients with:
* Chronic hypotension, systolic blood pressure < 100 mg Hg for women and < 110 mg Hg for men.
* Bradycardia, pulse < 50 beats per minute.
* Asthma or chronic obstructive lung disease
* Heart insufficiency with affected (< 50 %) left ventricle ejection fraction (LVEF), treated or untreated.
* Kidney insufficiency, defined as eGFR < 20 ml/min.
* Liver insufficiency defined as chronically high liver enzymes or known chronic liver disease (e.g., hepatitis, steatosis, cirrhosis).
* Cor pulmonale
* Cardiogenic shock
* Severe peripheral circulatory disorders
* Known or newly diagnosed current metabolic acidosis (e.g., in recent analysis of arterial puncture).
* Known hypersensitivity to propranolol or to one or more of the excipients.
* Currently untreated pheochromocytoma.
* History of Prinzmetals angina.
* History of sick sinus syndrome or atrioventricular block.
* History of stroke or any previous cardiovascular event.
* History of neoadjuvant oncological treatment for suspected primary pancreatic cancer.
* Recent or present (within 3 months) use of propranolol or any other beta-blocker.
* Recent or present (within 3 months) use of any of the following medications: anxiolytics, calcium channel blockers, beta-adrenergic receptor agonist.
* Medical history that classifies the patient as frail or unsuitable for inclusion by the examining physician.
* Histopathological examination revealing benign lesion.
* Predictable poor compliance, due to pre-existing psychiatric disease, dementia or not able to read or speak sufficient Danish, resulting in not being able to provide a well-informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Preoperative anxiety | Obtained preoperatively at baseline (immediately after inclusion) and immediately after intervention (before surgery)
  Assessed through the Hamilton Anxiety Rating Scale (HAMA) questionnaire
Preoperative anxiety and depression | Obtained preoperatively at baseline (immediately after inclusion) and immediately after intervention (before surgery)
  Assessed through the Hospital Anxiety and Depression Scale (HADS) questionnaire
Preoperative quality of life | Obtained preoperatively at baseline (immediately after inclusion) and immediately after intervention (before surgery)
  Preoperative quality of life assessed through the quality of life questionnaire.
Density and subtypes of tumor-infiltrating lymphocytes in the tumor microenvironment. | Through study completion. At latest within 1 year from last participant completes trial.
  Histopathological assessment of the density and subtypes of tumor-infiltrating lymphocytes.
  Immunohistochemistry technique will be used.
Desmoplasia in the tumor microenvironment. | Through study completion. At latest within 1 year from last participant completes trial.
  Histopathological assessment of desmoplasia in the tumor microenvironment.
  Immunohistochemistry technique will be used.
Neural markers in the tumor microenvironment. | Through study completion. At latest within 1 year from last participant completes trial.
  Histopathological assessment of neural marker expression (e.g., NGF, BDNF, tyrosin hydroxylase)
  Immunohistochemistry technique will be used.
Adrenergic receptor (ADRB1&ADRB2) expression in the tumor microenvironment. | Through study completion. At latest within 1 year from last participant completes trial.
  Histopathological assessment of the expression of adrenergic receptors (ADRB1 and ADRB2).
  Immunohistochemistry technique will be used for this purpose.
Spatial distribution of immune cells in the tumor microenvironment. | Through study completion. At latest within 1 year from last participant completes trial.
  Spatial distribution of immune cells in the tumor microenvironment using Immunohistochemistry technique and NanoString GeoMx techniques will be used for this purpose.
Immune cells and subtypes in blood samples | Through study completion. At latest within 1 year from last participant completes trial.
  Assessing the number and subsets of immune cells in the obtained blood samples before and after propranolol treatment and between the two arms (propranolol versus placebo). This will be examined through FlowCytometry.
Circulating tumor cells before and after intervention in blood samples. | Through study completion. At latest within 1 year from last participant completes trial.
  Assessment of circulating tumor cells in blood samples before and after intervention.
RNA-level gene expression in blood samples. | Through study completion. At latest within 1 year from last participant completes trial.
  RNA-level expression of genes related to immune-surveillance through NanoString nCounter technique.
Heart rate variability in both trial arms | Through study completion, an average of 1 year.
  Examining differences in heart rate variability among participants and between intervention and comparator group.
Postoperative complications | After participant finishes trial and when last follow up (5 years from surgery) date is due.
  Assessment of postoperative complications based on the Clavien-Dindo Score (CD) ranging from I to V, where I is any decline from normal postoperative course and V is death of patient.
Survival 30-days after surgery | After participant finishes trial and when last follow up (5 years from surgery) date is due.
  Assessment of survival 30 days after surgery.
Survival 90-days after surgery | After participant finishes trial and when last follow up (5 years from surgery) date is due.
  Assessment of survival 90 days after surgery.
Overall survival 1-year after surgery | After participant finishes trial and when last follow up (5 years from surgery) date is due.
  Assessment of overall surival 1-year after surgery
Overall survival 3-years after surgery | After participant finishes trial and when last follow up (5 years from surgery) date is due.
  Assessment of overall survival 3-years after surgery
Overall survival 5-years after surgery | After participant finishes trial and when last follow up (5 years from surgery) date is due.
  Assessment of overall survival 5-years after surgery

SECONDARY OUTCOMES:
Safety of 40 mg propranolol twice daily on blood pressure. | Through study completion, within 14 days after surgery.
  Examining the safety of preoperative propranolol 40 mg twice daily prior to elective surgery for pancreatic cancer by continuous at-home measurements of blood pressure twice daily during the intervention period.
Safety of 40 mg propranolol twice daily on heart rate. | Through study completion, within 14 days after surgery.
  Examining the safety of preoperative propranolol 40 mg twice daily prior to elective surgery for pancreatic cancer by continuous at-home measurements of heart rate twice daily during the intervention period.

OTHER OUTCOMES:
Feasibility of implementing preoperative propranolol in the preoperative setting for patients with pancreatic cancer using the APEASE framework. | Within 1 year from end of the trial.
  Examining the feasibility and implementation of preoperative 40 mg propranolol twice daily in patients undergoing surgery for pancreatic cancer. Challenges in the implementation will be assessed through the use of the APEASE framework, which looks in to Acceptability, Practicability, Effectiveness, Affordability, Spill-over effects, and Equity.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, Professor, Principal Investigator — Center for Surgical Science, Zealand University Hospital
Locations (2):
- Denmark (2):
  - Department of Surgical Gastroenterology, Copenhagen
  - Ismail Gögenur, Køge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Drug Information - Propranolol — https://dailymed.nlm.nih.gov/dailymed/search.cfm?labeltype=all&query=propranolol